CLINICAL TRIAL: NCT00731003
Title: The Effect of Serotonergic Modulation on Intestinal Permeability and Visceral Hypersensitivity in Healthy Individuals and IBS Patients
Brief Title: The Effect of Serotonergic Modulation on Intestinal Permeability and Visceral Hypersensitivity in Healthy Individuals and Irritable Bowel Syndrome (IBS) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MEC 08-2-070
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: serotonin; gut permeability; visceral sensitivity; irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — 5-Hydroxytryptophan; Tryptophan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- I (Experimental): ATD procedure
  Interventions: Other: Acute tryptophan depletion
- II (Experimental): Oxitriptan
  Interventions: Drug: Oxitriptan
- III (Placebo Comparator): Amino acid mixture with tryptophan
  Interventions: Other: Amino acid drink with tryptophan
- IV (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Oxitriptan — 100 mg 5-Hydroxytryptophan will be administered orally.
  Arms: II
Other: Acute tryptophan depletion — Acute tryptophan depletion employs the oral ingestion of an amino acid mixture devoid of tryptophan, the precursor of serotonin, which results in lowered serotonin levels.
  Arms: I
Other: Amino acid drink with tryptophan — Amino acid drink with tryptophan, placebo for the ATD procedure
  Arms: III
Drug: Placebo capsule — Placebo for 5-HTP
  Arms: IV

SUMMARY:
Serotonin, 5-hydroxytryptamin (5-HT), plays an important role in regulating the gastrointestinal functions. In this study we will modulate the serotonin system with acute tryptophan depletion (ATD) and administration of 5-hydroxytryptophan (5-HTP). ATD is based on ingestion of an amino acid drink devoid of the precursor of serotonin and hence caused a decreased serotonin level. 5-hydroxy-tryptophan is the direct precursor of serotonin and its administration, an increased serotonin level is expected. During these interventions, gut permeability and visceral sensitivity will be measured in healthy individuals and patients with irritable bowel syndrome, which is characterized by altered permeability and visceral hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* IBS-patients

Inclusion criteria:

1. IBS will be diagnosed according to the Rome III criteria* [35]:

   Recurrent abdominal pain or discomfort at least 3 days per month in the last 3 months associated with 2 or more of the following:
   * Improvement with defecation
   * Onset associated with a change in frequency of stool
   * Onset associated with a change in form (appearance) of stool

     * Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis
     * Discomfort means an uncomfortable sensation not described as pain. In pathophysiological research and clinical trails, a pain/discomfort frequency of at least 2 days a week during screening evaluation is an indication for subject's eligibility.
2. Based on the medical history and previous examination, no other causes for the abdominal complaints can be defined.
3. Age between 18 and 65 years

Healthy individuals

Inclusion criteria:

All subjects will be screened with a standardized psychiatric examination using the mini international neuropsychiatric interview (MINI) to determine present psychiatric state. General psychological state will be assessed using the 17 item Hamilton depression rating scale (HAM-D17), the Dutch version of the symptom checklist (SCL-90) and the hospital anxiety and depression rating scale (HADS). The psychiatric evaluation will be carried out by a psychiatrist. Volunteers with deviating scores on any topic will be excluded from participation.

Healthy individuals between age 18 and 65 years will be included in the study.

Exclusion Criteria:

* Exclusion criteria for IBS patients:

  1. Severe co-morbidity hindering a rectal barostat procedure, according to the gastroenterologist's perception.
  2. Abdominal surgery, except for uncomplicated appendectomy, laparoscopic cholecystectomy or hysterectomy.
  3. Inability to stop medication that can influence gastrointestinal motility or perception (like loperamide, butylscopolamine, psylliumsead (metamucil), duspatal, metoclopramide, domperidon, erytromycine), or serotonin metabolism (carbidopa) for at least 3 days before tests.
  4. History of psychiatric disorders including use of psychoactive medication or psychological symptomatology, defined as a diagnosis on the MINI, HAM-D17 score above 18, global severity index score on SCL-90 for females ≥150, for males ≥131, or HADS scores ≥ 8. First-degree family members with psychiatric disorders
  5. Administration of investigational drugs in the 180 days prior to the study
  6. Premenstrual syndrome, dieting, pregnancy, lactation
  7. Excessive alcohol consumption (>20 alcoholic consumption per week)
  8. Smoking
  9. Blood donation within 3 months before the study period
  10. Self-admitted HIV-positive state
  11. Irregular day-night rhythm

Exclusion criteria for healthy individuals:

1. History of gastrointestinal, psychiatric disorders including use of psychoactive medication or psychological symptomatology, defined as a diagnosis on the MINI, HAM-D17 score above 18, global severity index score on SCL-90 for females ≥150, for males ≥131, or HADS scores ≥ 8 First-degree family members with psychiatric disorders
2. Use of medication, except oral contraceptives, within 14 days prior to testing
3. Administration of investigational drugs in the 180 days prior to the study
4. Previous abdominal surgery (other than uncomplicated appendectomy, laparoscopic cholecystectomy and hysterectomy)
5. Premenstrual syndrome, dieting, pregnancy, lactation
6. Excessive alcohol consumption (>20 alcoholic consumption per week)
7. Smoking
8. Blood donation within 3 months before the study period
9. Self-admitted HIV-positive state
10. Irregular day-night rhythm
11. Severe co-morbidity hindering a rectal barostat procedure, according to the gastroenterologist's perception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary aim is to assess intestinal permeability under altered serotonergic conditions by means of sugar permeability test | 2010

SECONDARY OUTCOMES:
To assess tight junction functionality and serotonin metabolism To assess visceral hypersensitivity under altered serotoninergic conditions To examine biopsy specimens for serotonergic and intestinal permeability parameters in ex vivo circumstances | 2010

CONTACTS AND LOCATIONS:
Overall Officials: A AM Masclee, Prof. Dr., Principal Investigator — Maastricht University Hospital; F Troost, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

REFERENCES:
- [Result] Keszthelyi D, Troost FJ, Jonkers DM, van Eijk HM, Lindsey PJ, Dekker J, Buurman WA, Masclee AA. Serotonergic reinforcement of intestinal barrier function is impaired in irritable bowel syndrome. Aliment Pharmacol Ther. 2014 Aug;40(4):392-402. doi: 10.1111/apt.12842. Epub 2014 Jun 18. PMID 24943480
- [Result] Keszthelyi D, Troost FJ, Jonkers DM, Kruimel JW, Leue C, Masclee AA. Decreased levels of kynurenic acid in the intestinal mucosa of IBS patients: relation to serotonin and psychological state. J Psychosom Res. 2013 Jun;74(6):501-4. doi: 10.1016/j.jpsychores.2013.01.008. Epub 2013 Feb 15. PMID 23731747
- [Result] Keszthelyi D, Troost FJ, Jonkers DM, van Donkelaar EL, Dekker J, Buurman WA, Masclee AA. Does acute tryptophan depletion affect peripheral serotonin metabolism in the intestine? Am J Clin Nutr. 2012 Mar;95(3):603-8. doi: 10.3945/ajcn.111.028589. Epub 2012 Feb 1. PMID 22301931